CLINICAL TRIAL: NCT04386031
Title: Fungal Infection After Oral Cavity Surgeries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0196-19-RMB CTIL
Record Dates: First submitted 2020-05-10; First posted 2020-05-13 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Prevalence of Fungal Infection in Patients Undergoing Oral Cavity Surgery Without Treatment With Antifungal Drug

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- group with antifungal drug
  Interventions: Diagnostic Test: Throat culture for fungal pathogens
- A control group: A control group will be taken ,patients undergoing thyroidectomy or parotidectomy
  Interventions: Diagnostic Test: Throat culture for fungal pathogens

INTERVENTIONS:
Diagnostic Test: Throat culture for fungal pathogens — Throat culture for fungal pathogens will be taken before surgery, at post-operative day (POD) 3 and 2 weeks after the operation

SUMMARY:
this prospective study we will examine the prevalence of fungal infection in patients undergoing oral cavity surgery without treatment with antifungal drug

ELIGIBILITY:
Inclusion Criteria:

* Age over 18

Exclusion Criteria:

* Previous oral cavity surgery.

  * Previous radiotherapy to the head and neck.
  * Previous treatment with antifungal drugs in the 30 days preceding the surgery Immunocompomised state at the date of surgery.
  * Pregnancy
  * Lack of follow-up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years old, undergoing oral cavity surgery at ENT department and maxillofacial surgery department, Rambam medical center between May 2019-May 2021
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of fungal infection in patients undergoing oral cavity surgery without treatment with antifungal drug. | 2 years
  40 patients undergoing oral cavity surgery and 40 patients (control group) undergoing thyroidectomy or parotidectomy for our research measurement :Throat culture for fungal pathogens